CLINICAL TRIAL: NCT07101861
Title: Breast Cancer Survivors RESET (Reducing Weight and Elevated Stress Levels Using Educational and Behavioral Tools): A Pilot, Feasibility Study
Acronym: RESET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: MCC-22616
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survivors RESET intervention (Experimental)
  Interventions: Behavioral: Survivors RESET

INTERVENTIONS:
Behavioral: Survivors RESET — 16-session adaptation of the Diabetes Prevention Program Intensive Lifestyle Intervention plus stress management training

SUMMARY:
The overall object of this project is to test the feasibility and acceptability of an adapted stress management enhanced behavioral weight loss intervention for Black breast cancer survivors with obesity and elevated stress. We will also conduct pre- and post-intervention assessments of weight, allostatic load, and patient reported outcomes among study participants.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as non-Hispanic Black
* Self-identify as cisgendered female.
* Are ≥ age 18.
* Have a history of stage 0-3 breast cancer diagnosis treated for curative intent.
* Have completed all adjuvant or neoadjuvant chemotherapy, radiation, and surgery at least 21 days prior to study registration but may continue on hormonal therapy and Abemaciclib therapy.
* Have a measured BMI ≥ 30 kg/m2.
* Willing to participate for the entire 4-month duration.

Exclusion Criteria:

* Are pregnant or are planning to become pregnant during the study period.
* Have a known major medical or psychological condition known to influence weight loss [e.g., medicated or poorly controlled diabetes (HbA1c > 8%), uncontrolled hypertension (BP>160 mm Hg systolic or BP>100 mm Hg diastolic), cardiovascular event in the past 12 months, history of gastric bypass or bariatric surgery].
* History of psychiatric hospitalization in past 2 years.
* History of substance abuse or eating disorder.
* Any other condition by which a medical professional has suggested diet modification, physical activity, and/or weight loss would be contraindicated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Enrollment Rate | Baseline
  Percentage of participants who are contacted and enroll in the study.
Retention Rate | Baseline to Month 4
  Percentage of participants who enroll and complete assessments at both timepoints (Baseline and Month 4).
Adherence | Baseline to Month 4
  Adherence will be assessed by the number of treatment sessions attended.

SECONDARY OUTCOMES:
4-month mean change in weight | Baseline to Month 4
  Weight change as measured by a SECA scale in kilograms at baseline and month 4 will be calculated and averaged
4-month mean change in allostatic load score | Baseline to Month 4
  Allostatic load score will be calculated using a validated equation. Change from baseline to month 4 will be calculated and averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Carson, PhD, MPH, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States